CLINICAL TRIAL: NCT03319472
Title: Clinical Identification of Malignant Pleural Effusions in the Emergency Department
Brief Title: Using Pleural Effusions to Diagnose Cancer
Acronym: MAPED
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Georgios Stathopoulos, Associate Professor of Physiology, University of Patras
Other Study IDs: 22699/21.11.2013
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Pleural Effusion
Keywords: malignant; cancer; simple bedside test; rapid; score; widely available; feasible
MeSH Terms: conditions — Pleural Effusion; Neoplasms; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pleural fluid will be centrifuged and cells will be separated from supernatants. The latter will be stored together with matched serum samples at -80 degrees C. Cell pellets will be stored in DMEM 10% FBS, 2 % DMSO at the same temperature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign Pleural Effusion: Patients that will be diagnosed within a month from admission with any non-malignant cause of pleural effusion, including but not limited to effusions caused by common or tuberculous or fungal infection, heart failure, etc. Documentation of the etiology will be required for inclusion in this group, including but not limited to bacteriology, virology, PCR, radiology, heart echocardiogram or catheterization, as appropriate.
- Malignant Pleural Effusion: Patients that will be diagnosed within a month from admission with any malignant cause of pleural effusion, including but not limited to effusions caused by lung, breast, colon, ovary, mesothelial, hematopoietic, prostate, or any other cancer. Diagnosis will be based on verification of the presence of malignant cells in the pleural fluid or tissues. Patients with cancer and an effusion without such documentation will be assigned to the benign group if an alternative diagnosis is made. In any other case, they will be excluded.

SUMMARY:
Pleural effusions (PE) are common conditions that signal either infection or cancer. The investigators aim to develop, validate, and prospectively assess the MAPED score, a clinical score that predicts malignancy at admission. This tool will assist clinicians all over the world to rapidly assess the probability of an effusion being malignant within 4 hours of admission.

DETAILED DESCRIPTION:
Background: Pleural effusions (PE) are common conditions that signal either pleural-disseminated infection or cancer. While these diagnoses bear tremendous importance for patients, they require invasive procurement of pleural tissues and/or cells and time. Simple and rapid diagnostic markers of pleural malignancy at admission that streamline diagnostic and treatment efforts remain unidentified.

Objective: To develop, validate, and prospectively assess markers of malignancy of PE at admission.

Methods: A prospective cohort of patients with PE from different etiologies will be recruited stating on 11.21.2013 and prospectively ending on 11.21.2023. Data will be collected within 4 hours of admission including history, chest X-ray, and blood and pleural fluid (PF) cell counts and basic biochemistry. Pleural fluid and serum will be biobanked for future analyses. Patients will sign informed consent forms. Diagnosis will be confirmed using standard microbiology, cytology, histology, and imaging techniques. Patients undiagnosed within a month will be excluded. Variables will be entered into binary regression and receiver-operator analyses using malignancy as the target to develop the MAPED score, a clinical score that predicts malignancy at admission. MAPED will be retrospectively validated in separate published cohorts from the first therapeutic interventions in malignant effusion (TIME) 1-3 trials from Oxford UK. Data will be censored and analyzed three times, at 40-month intervals since study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Pleural effusion
* Hospital admission
* No previous pleural procedure
* Age > 18 years
* No previous chemoradiotherapy
* No antibiotic therapy during previous trimester
* All history, chest X-ray, and pleural and blood cell counts and biochemistry entry data obtained within 4 hours after admission

Exclusion Criteria:

* No diagnosis at one month post-admission
* No informed consent provided
* Age < 18 years
* History, chest X-ray, or pleural and blood cell counts and biochemistry entry data obtained later than 4 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to a tertiary hospital with a pleural effusion.
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Malignancy | One month post-admission
  Cytologic or histologic evidence of malignant cells or tissues in the pleural space.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios T Stathopoulos, MD, PhD, Principal Investigator — Associate Professor of Physiology
Locations (1):
- Patras University Hospital, Rio, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Undecided